CLINICAL TRIAL: NCT02031848
Title: Brain Function Predictors And Outcome Of Weight Loss And Weight Loss Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cary Savage, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Cary Savage, Ph.D., Director, CHBN and John H. Wineinger Professor of Psychiatry and Behavioral Sciences, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11123
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Obesity
Keywords: weight loss; diet
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Weight Control Group (Active Comparator): Subjects will complete the Assessments, Diet Intake, and MRI portions of the study
  Interventions: Other: Assessments and Diet Intake
- Dieting Group (Active Comparator): Subjects will complete the Assessments, Diet Intake, and MRI portions of the study and will be given the weight loss and weight maintenance diets, and will attend weekly behavioral meetings
  Interventions: Other: Diet Intervention

INTERVENTIONS:
Other: Diet Intervention
  Arms: Dieting Group
Other: Assessments and Diet Intake
  Arms: Healthy Weight Control Group

SUMMARY:
By doing this study, researchers hope to learn whether a person's motivation for food is different after he or she loses weight, and if imaging techniques such as fMRI can be used to predict whether the person will maintain that weight loss over time.

ELIGIBILITY:
Inclusion Criteria:

* BMI equal to or greater than 30 kg/m2 or 18 to 24.9
* declaration they do not have plans to move out of the Greater Kansas City area for at least 1 year
* willingness to be randomized
* Individuals undergoing weight loss will have to present written approval from a licensed physician that they are healthy enough to participate in a program of moderate diet restriction and moderate physical activity.

Exclusion Criteria:

* Participation in a research project involving weight loss or PA in the previous 6 months, as these proximal experiences may impact the results of this study.
* Subjects who smoke
* Subjects who use special diets (i.e. vegetarian, Adkins, etc.), use medications that affect metabolism (i.e. thyroid, beta blockers), use medications that affect appetite (i.e. Meridia) or cannot exercise (i.e. walk).
* Exhibit signs of eating disorders, restraint, depression
* Participant has any metabolic disease that would affect energy balance (e.g. diabetes mellitus or hypothyroidism).
* Individuals who report being pregnant during the previous 6 months, are lactating, or planned pregnancy within 12 months
* Individuals who are not weight stable (± 4.5kg) within the previous 3 months or have more than 500 kcal/wk of planned physical activity
* Serious medical risk such as type 1 diabetes, cancer, recent cardiac event (i.e. heart attack, angioplasty, etc.)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2008-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Differences in brain activation to visual food cues | Change from Baseline to 3 Months
  differences will be measured by scanning subjects with fMRI and measuring changes in different regions of the brain.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kansas, Lawrence, Kansas

REFERENCES:
- [Derived] Honea RA, Szabo-Reed AN, Lepping RJ, Perea R, Breslin F, Martin LE, Brooks WM, Donnelly JE, Savage CR. Voxel-based morphometry reveals brain gray matter volume changes in successful dieters. Obesity (Silver Spring). 2016 Sep;24(9):1842-8. doi: 10.1002/oby.21551. Epub 2016 Jul 19. PMID 27430417
- [Derived] Szabo-Reed AN, Breslin FJ, Lynch AM, Patrician TM, Martin LE, Lepping RJ, Powell JN, Yeh HW, Befort CA, Sullivan D, Gibson C, Washburn R, Donnelly JE, Savage CR. Brain function predictors and outcome of weight loss and weight loss maintenance. Contemp Clin Trials. 2015 Jan;40:218-31. doi: 10.1016/j.cct.2014.12.008. Epub 2014 Dec 19. PMID 25533729